CLINICAL TRIAL: NCT05613803
Title: The Efficacy and Mechanisms of Action of n-3 Poly-unsaturated Fatty Acid Supplementation in People With Non-steroidal Exacerbated Airways Disease and Uncontrolled Asthma
Brief Title: Poly-unsaturated Fats for Improving Nasal Polyps and Asthma
Acronym: PUFFIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (173-12-20)
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish oil (Active Comparator): 6g of Eicosapentaenoic acid (EPA) and Docosahexaenoic acid (DHA) in a 1.3:1 ratio; respectively, as six Omacor capsules, taken once daily, or in divided doses, with food.
  Interventions: Drug: Fish oil
- Placebo (Placebo Comparator): Matched capsules (six) containing palm olein IV 56 taken once daily, or in divided doses, with food.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fish oil — 6g of EPA and DHA in a 1.3:1 ratio as six Omacor capsules manufactured by Provona Biocare (Olso Norway), or generic equivalent, taken once daily, or in divided doses, with food.
  Other Names: Active arm
  Arms: Fish oil
Other: Placebo — Six capsules containing palm oil and soybean oil on an 8:2 ratio taken once daily, or in divided doses, with food.
  Other Names: Control arm
  Arms: Placebo

SUMMARY:
Asthma is a syndrome compromising many phenotypes including N-ERD (caused by increased 4-series leukotriene (LT) production). n-3 PUFA supplementation modulates 4-series LT and has anti-inflammatory effects. However, other than in a pilot study with dietary manipulation, the effects of N-ERD are unknown. The primary objective is to determine whether n-3 PUFA supplementation in people with N-ERD can improve asthma control using the asthma control questionnaire (ACQ-7). This is a placebo controlled randomised controlled parallel multicentre study with of 6g per day of PUFA for 6 months in people with N-ERD and poor asthma control

DETAILED DESCRIPTION:
Asthma is a syndrome compromising many phenotypes including N-ERD (caused by increased 4-series leukotriene (LT) production). n-3 PUFA supplementation modulates 4-series LT and has anti-inflammatory effects. However, other than in a pilot study with dietary manipulation, the effects of NERD are unknown.

The primary objective is to determine whether n-3 PUFA supplementation in people with N-ERD can improve asthma control using the asthma control questionnaire (ACQ-7). Secondary objectives are to determine whether n-3 PUFA improves asthma and rhinitis symptoms and quality of life and airway calibre. Mechanistic objectives are to assess effects on red blood cell fatty acid composition, cyclooxygenase pathways and airway inflammation.

This is a placebo controlled randomised controlled parallel multicentre study with of 6g per day of PUFA for 6 months in people with N-ERD and poor asthma control. Ninety-eight people will be included in the study if they have a reliable history of N-ERD or a positive nasal aspirin challenge, an ACQ-7 > 1.5 and are on stable treatment. People with other significant disease, recent respiratory tract infection, receiving aspirin desensitisation, biological asthma therapies will be excluded, as will those with a significant smoking history or alcohol consumption. The intervention will be 6g of n-3 PUFA (EPA and DHA as six (5.04g EPA+DHA) taken once daily, or in divided doses, with food for 6 months. The control will be matched placebo. Measurements will be at be made at baseline, 3 months and 6 months for ACQ-7 (equivalent to ACQ-6 plus spirometry), exhaled nitric oxide (FeNO) and blood for red blood cell fatty acid concentration, blood eosinophil count and safety markers. The following questionnaires will also be undertaken at these time-points: Mini Asthma Quality of Life Questionnaire (mini-AQLQ), and Euroqol 5 dimension 5 level (EQ5D-5L). The ACQ-6 will be measured every 6 weeks throughout the study and the food frequency questionnaire will be measured at baseline and 6 months. Urine will be analysed for uLTE4 and prostaglandin D2 at baseline and 6 months. Induced sputum will be obtained at baseline and 6 months in a subgroup for differential cell count and specialised pro-resolving mediators.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years. N-ERD does not occur at birth and it rarely occurs in children.
2. physician labelled diagnosis of asthma.
3. history of N-ERD according EAACI guidelines(9) with evidence of one of 1) Clinical diagnosis as evidence by i. A reliable history of aspirin or NSAID induced respiratory reaction as evidenced by more than one reaction, reactions to two or more different NSAIDs or the last reaction occurring within the last 5 years plus ii. Recurrent nasal polyposis, anosmia, moderate to severe asthma, intolerance to alcohol and/or blood eosinophilia 2) Positive nasal or bronchial aspirin challenge(43)
4. ACQ of more than 1.5 as this indicates poor control. This is required to ensure there is a clinical need or a requirement to alter medication.
5. stable disease, as evidenced by a lack of change in asthma therapy within the last 6 weeks.

Exclusion Criteria:

1. significant cardiac disease, respiratory disease or other cause for breathlessness other than asthma
2. severe or uncontrolled co-morbid disease (other than nasal polyps) which is likely to affect the outcome of the study
3. having had an upper or lower respiratory tract infection requiring antibiotics within four weeks of randomisation
4. receiving aspirin desensitisation therapy or biologic agents
5. receiving n-3 fatty acid oral supplements
6. current smoker or more than 15 pack-year smoking history
7. consumption of more than 21 units of alcohol per week as alcohol-induced respiratory symptoms are more common in N-ERD.
8. patients unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Questionnaire (ACQ) 6 | 24 weeks post-randomisation
  Asthma control questionnaire (ACQ) mean score of more than 1.5, as this indicates poor control. This is required to ensure there is a clinical need or a requirement to alter medication.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilson, Principal Investigator — University of East Anglia
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom